CLINICAL TRIAL: NCT03978156
Title: Dronabinol for Pain and Inflammation in Adults Living With Sickle Cell Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Covid-19. Relocation of trainee/investigator. Covid-19.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000021179
Record Dates: First submitted 2019-05-22; First posted 2019-06-06 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Dronabinol; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blind, cross-over study of dronabinol compared to placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dronabinol, Then Placebo (Experimental): Participants will take 2.5 mg of Dronabinol for 2 weeks, 1 week washout and then take 2 weeks of placebo (microcrystalline cellulos). Subjects will take up to 8 capsules daily of the treatment daily during each phase.
  Interventions: Drug: Dronabinol 2.5 MG; Drug: Microcrystalline cellulose
- Placebo, Then Dronabinol (Experimental): Participants will take placebo (microcrystalline cellulos) for 2 weeks, 1 week washout and then take 2.5 mg of Dronabinol for 2 weeks. Subjects will take up to 8 capsules daily of the treatment daily during each phase.
  Interventions: Drug: Dronabinol 2.5 MG; Drug: Microcrystalline cellulose

INTERVENTIONS:
Drug: Dronabinol 2.5 MG — Subjects will take dronabinol daily during 2 week dosing period separated by a one week washout period.
Drug: Microcrystalline cellulose — Subjects will take placebo daily during 2 week dosing period separated by a one week washout period.
  Other Names: Placebo

SUMMARY:
This study is designed to address the feasibility of a randomized, double masked, cross-over study of dronabinol as a palliative agent in the treatment of pain, inflammation, and other complications of sickle cell disease (SCD).

DETAILED DESCRIPTION:
The Primary Hypothesis is that such a study will be feasible as defined by subject adherence to study medication and study procedures and avoidance of other cannabinoid containing substances during the trial period as well as by ability to mask subjects and investigators to treatment assignment

Secondary hypotheses are:

Dronabinol will:

Reduce patient-reported pain interference Reduce patient-reported pain scores and change patient-reported pain quality. Reduce use of opioid pain medications. Improve patient-reported stiffness, nausea and vomiting, sleep, mood, anxiety, and social functioning.

Reduce markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥18 years, able to understand and sign the informed consent form
* Clinical diagnosis of SCD (HbSS, HbSC, HbSβ+; Thal, HbSβ0Thal, HbS variants)
* Baseline score of 60 or lower on the ASCQ-Me 7-day pain interference domain
* Willing to abstain from marijuana, medical and illicit, during study weeks 1 through 6.
* For patients currently receiving hydroxyurea and/or L-glutamine, on a stable dose(s) for at least 3 months
* For patients currently on a chronic red blood cell transfusion program, on such a program for at least 3 months

Exclusion Criteria:

* Known intolerance to dronabinol, sesame oil, or marijuana
* Patients with a diagnosis or medical history of any psychiatric disorder with psychosis
* Presence of any concomitant medical condition, or use of concomitant medication, that, in the Investigator's opinion, may place the subject at increased risk of side effects of dronabinol.
* Pregnant or nursing women
* If a woman capable of becoming pregnant, unwilling to use a medically accepted form of birth control for the duration of study participation. Accepted forms include oral contraception or vaginal ring, medroxyprogesterone, contraceptive implants, intrauterine device, or patch, surgical sterilization, total abstinence. We have not included a similar restriction for men as the current FDA approval includes no such restriction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Feasibility will be defined by ability to mask patients and investigators to treatment assignment and adherence | 1 year
  Feasibility will be defined by ability to mask patients and investigators to treatment assignment and adherence which will be defined in 3 ways.
Adherence | 1 year
  Adherence to study drug will be assessed with weekly pill counts and urine toxicology.
Avoidance | 7 weeks
  Avoidance of other cannabinoid containing substances will also be defined using urine toxicology once at the end of each treatment period and once at the end of the wash out period.
Adherence to other study proceedures | 7 weeks
  Adherence to other study procedures will be defined as percent of visits attended, percent of urine and serum studies collected and percent of patient reported outcomes and daily pain severity and pain unpleasentness journals returned.

SECONDARY OUTCOMES:
Patient reported 7-day pain interference | 7 days
  The primary endpoint for this study will be second treatment week 7-day pain impact as measured by the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) 7-day pain impact domain. ASCQ-Me domains are validated to measure pain and other quality of life outcomes in adults with Sickle Cell Disease (SCD) of all genotypes. The published mean for the validated scores is 50 and the standard deviation is 10.56 Lower scores represent more severe symptoms. When the validation cohort was placed into tertiles of severity, the tertile with most severe disease had a mean pain score of 53, the middle tertile had a score of 49, and the least severe disease tertile had a mean score of 46. This suggests that a change of 4 has clinical significance and a change of 7 has even more clinical significance. We have chosen a priori to define a difference in pain impact score of 5 points as showing superiority.
Patient Pain Severity | end of 2nd week
  Daily reports of pain severity on a numeric rating scale of 0-10 with 0 representing the least severe pain (no pain) and 10 representing the most severe pain.
Patient Pain Unpleasantness | end of 2nd week
  Daily reports of pain unpleasantness on a numeric rating scale of 0-10 with 0 representing the least pain unpleasantness (no unpleasantness) and 10 representing the most unpleasant pain.
PROMIS (Patient Reported Outcomes Measurement Information System) Nociceptive Pain Severity | end of 2nd week
  Nociceptive pain quality as defined by the patient report outcome measurement information system (PROMIS) nociceptive pain quality 5a scale. All PROMIS scores will be presented as T scores. The T score is a standardized score with a mean of 50 and a standard deviation of 10. The value of 50 represents the score of the average field test respondent.
PROMIS Neuropathic Pain Severity | end of 2nd week
  Neuropathic pain quality as defined by the patient report outcome measurement information system (PROMIS) neuropathic pain quality 5a scale.All PROMIS scores will be presented as T scores. The T score is a standardized score with a mean of 50 and a standard deviation of 10. The value of 50 represents the score of the average field test respondent.
PROMIS Gastrointestinal Nausea short form measure | end of 2nd week
  PROMIS short form Gastrointestinal Nausea and vomiting 4a. All PROMIS scores will be presented as T scores. The T score is a standardized score with a mean of 50 and a standard deviation of 10. The value of 50 represents the score of the average field test respondent.
PROMIS short form for emotional distress anxiety 8a. | end of 2nd week
  PROMIS short form Gastrointestinal Nausea and vomiting 4a. All PROMIS scores will be presented as T scores. The T score is a standardized score with a mean of 50 and a standard deviation of 10. The value of 50 represents the score of the average field test respondent.
Adult Sickle Cell Quality (ASCQ)-Me short form measures of emotional impact | end of 2nd week
  Each ASCQ-Me score is reported on the same standardized scale with a mean of 50 and a standard deviation of 10. The value of 50 represents the health score of the average field test respondent.
Adult Sickle Cell Quality (ASCQ)-Me short form measure of sleep impact | end of 2nd week
  Each ASCQ-Me score is reported on the same standardized scale with a mean of 50 and a standard deviation of 10. The value of 50 represents the health score of the average field test respondent.
Adult Sickle Cell Quality (ASCQ)-Me short form measure of stiffness impact | end of 2nd week
  Each ASCQ-Me score is reported on the same standardized scale with a mean of 50 and a standard deviation of 10. The value of 50 represents the health score of the average field test respondent.
Adult Sickle Cell Quality (ASCQ)-Me short form measure of social functioning impact | end of 2nd week
  Each ASCQ-Me score is reported on the same standardized scale with a mean of 50 and a standard deviation of 10. The value of 50 represents the health score of the average field test respondent.
Opioid Utilization | end of 2nd week
  Secondary comparisons will be made between subjects on dronabinol to themselves on placebo for patient reported outcomes for opioid use. Opioid utilization will be based on reports of opioids dispensed obtained from the Connecticut Prescription Monitoring Program. Reports will be in the form of average daily opioids used in oral morphine equivalents.
Markers of Inflammation Concentration of white blood cell count differential | end of 2nd week
  Secondary comparisons will be made between subjects on dronabinol to themselves on placebo for differential white blood cell count at the end of the second week of the treatment period.
Markers of Inflammation C reactive protein | end of 2nd week
  Secondary comparisons will be made between subjects on dronabinol to themselves on placebo of C reactive protein at the end of the second week of the treatment period.
Markers of Inflammation serum tryptase | end of 2nd week
  Secondary comparisons will be made between subjects on dronabinol to themselves on placebo for serum tryptase at the end of the second week of the treatment period.
Serum pro-inflammatory cytokines | end of 2nd week
  Secondary comparisons will be made between subjects on dronabinol to themselves on placebo for pro-inflammatory cytokines at the end of the second week of the treatment period.
Serum measure of Substance P | end of 2nd week
  Secondary comparisons will be made between subjects on dronabinol to themselves on placebo for Substance P at the end of the second week of the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Curtis, MD, Principal Investigator — Yale University School of Medicine Oncology Section
Locations (1):
- Yale New Haven Hospital Smilow Cancer Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Curtis SA, Jhawar R, Bellis J, McCuskee S, Devine L, Roberts JD. A pilot study of dronabinol for the treatment of pain in sickle cell disease. Pilot Feasibility Stud. 2025 Nov 12;11(1):139. doi: 10.1186/s40814-025-01705-6. PMID 41225660